CLINICAL TRIAL: NCT04507412
Title: Effect of Perioperative Intravenous Dexamethasone Administration in Patients Undergoing Total Shoulder Arthroplasty for Osteoarthritis, in Terms of Post-operative Pain, Function, Nausea, Hospitalization Length, and Risk of Complications
Brief Title: Intravenous Dexamethasone Administration in Patients Undergoing Total Shoulder Arthroplasty
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Christian Candrian (Other)
Responsible Party: Sponsor-Investigator, Christian Candrian, Principal Investigator, Ente Ospedaliero Cantonale, Bellinzona
Organization: Ente Ospedaliero Cantonale, Bellinzona (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ORL-ORT- 020
Record Dates: First submitted 2020-08-07; First posted 2020-08-11 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Arthroplasty, Replacement, Shoulder
Keywords: Total Shoulder Arthroplasty; steroid
MeSH Terms: interventions — Dexamethasone; Steroids

STUDY DESIGN:
Intervention Model Description: This study is a 2-arm randomized controlled trial comparing i.v. dexamethasone supplementation (arm-A) and no steroid supplementation (arm-B) for total shoulder arthroplasty
Who Masked: Participant, Outcomes Assessor
Masking Description: The present study will be double blinded: both participants and assessors will be blinded to the assigned treatment. Surgeons will be also blinded, only anaesthetists taking part to surgery will be aware of the group to which the patient was assigned but they will not take part to the follow-up visits.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- arm A (Experimental): • 9 mg of i.v. dexamethasone
  Interventions: Drug: dexamethasone
- arm B (No Intervention): • no steroid supplementation

INTERVENTIONS:
Drug: dexamethasone — perioperatively 9 mg i.v subministration
  Other Names: Steroids
  Arms: arm A

SUMMARY:
The aim of the study is to evaluate if intravenous steroid supplementation can provide advantages over routine analgesia protocols in terms of post-operative symptoms (pain and nausea), length of hospital stay, shoulder range of motion, function and patient satisfaction

DETAILED DESCRIPTION:
The purpose of this study is to detect the efficacy of intravenous perioperative steroid supplementation for total shoulder arthroplasty (TSA) surgeries in terms of short-term and long-term clinical outcomes and to demonstrate its advantages over the routine anaesthesia protocol. The comparison will be evaluated in terms of post- operative pain and function, opioids and analgesic drugs consumption, patient satisfaction, patient reported outcome measures (validated clinical scores), clinician-assessed clinical scores, systemic inflammatory response, length of hospital stay and long-term outcomes. Moreover, to confirm the safety of steroid supplementation all treatment related adverse events- and reactions are going to be recorded and reported, as well as post-operative glycaemia will be monitored.

The primary objective of the study is to show the efficacy on post-operative pain of intravenous perioperative dexamethasone supplementation for TSA.

The secondary objectives of the study are to show superiority by comparison of the intravenous peri- operative dexamethasone supplementation group to the routine analgesia protocol (no steroid supplementation group), in terms of post-operative pain and function, patient satisfaction, shoulder active- and passive range of motion, quantification with validated clinician- and patient reported outcome measures as the Constant, ASES and SSV Scores for function and EQ-5D-3L Score for health-related quality of life, opioids and analgesic drugs consumption, systemic inflammatory response, time until first mobilization and until the patient first slept through at night, the length of hospital stay and presence or absence of a frozen shoulder at the postoperative follow-up, as well as adverse events and reactions, in order to document the advantage over the absence of steroid supplementation in the short-, mid- term- and long-term follow up.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing unilateral primary total anatomical or reverse shoulder arthroplasty (Total Shoulder Arthroplasty)
* Patients with a BMI >18.5 and <35
* Patients able to provide informed consent and follow all the study procedures as indicated by the protocol
* Informed Consent as documented by signature

Exclusion Criteria:

* Contraindications to steroids
* Revision and post-traumatic TSA
* Active steroid or immunosuppressive therapy in the last 30 days before the operation
* Pregnant or breast-feeding women
* Presence of other clinically significant concomitant disease states (ASA IV)
* Uncontrolled diabetes mellitus
* Contraindications to Non-steroidal anti-inflammatory drugs
* Chronic systemic diseases as immunodeficiency, autoimmune disease (Systemic Lupus Erythematosus), gout, rheumatic arthritis
* Known or suspected non-compliance, drug or alcohol abuse
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant.
* Participation in another study with investigational drug within the 30 days preceding and during the present study
* Previous enrolment into the current study
* Enrolment of the investigator, his/her family members, employees and other dependent persons

Ages: 58 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2020-09-09 (Actual); Primary Completion 2032-07-31 (Estimated); Study Completion 2032-08-31 (Estimated)

PRIMARY OUTCOMES:
mean post-operative daily pain at rest | first 3 days after surgery
  0-10 numeric rating scale (NRS)from 0 to 10, with 10 being most painful

SECONDARY OUTCOMES:
Post-operative shoulder pain | first 3 months after surgery
  0-10 numeric rating scale (NRS)from 0 to 10, with 10 being most painful
Post-operative shoulder pain | 2 and 6 weeks after surgery and 3, 6, 12, 24, 60 ,120 months after surgery
  0-10 numeric rating scale (NRS)from 0 to 10, with 10 being most painful
Post-operative global shoulder function score | daily during the first 3 months
  0-10 numeric rating scale (NRS)from 0 to 10, with 10 being most functional
Post-operative global shoulder function score | 2 and 6 weeks after surgery and 3, 6, 12, 24, 60 ,120 months after surgery
  0-10 numeric rating scale (NRS)from 0 to 10, with 10 being most functional
The clinician assessed Constant score | 2 and 6 weeks after surgery and 3, 6, 12, 24, 60 ,120 months after surgery
  The Constant Score questionnaire consists of 8 questions (giving a score of 0 -100, with 100 being the best score) evaluating pain, activity level and range of motion
The American Shoulder and Elbow Surgeons Standardized Shoulder Assessment Form (ASES Score) | 2 and 6 weeks after surgery and 3, 6, 12, 24, 60 ,120 months after surgery
  The ASES Score is a patient reported outcome measure (PROM), a validated score evaluating pain and function for daily living and leisure activity. A maximum of 100 points means maximum (normal) functionality and no pain. MCID is 13.6 ± 2.3 points after total shoulder prosthesis
The Subjective Shoulder Value (SSV) | 2 and 6 weeks after surgery and 3, 6, 12, 24, 60 ,120 months after surgery
  The SSV is a percent of the subjective value of the shoulder given from the patient from 0-100%.
European Quality of Life-5 Dimensions-3 Level | 2 and 6 weeks after surgery and 3, 6, 12, 24, 60 ,120 months after surgery
  "Health-Related Quality-of-Life Score" and is preferred evaluating cost utility analysis and changes in general health after surgical operations. It contains 5 questions and the maximum (best) score is 1. MCID is 0.07 units
PainDETECT | 2 and 6 weeks after surgery and 3, 6, 12, 24, 60 ,120 months after surgery
  PainDETECT consists of seven questions that address the quality of pain symptoms; it is completed by the patient and no physical examination is required. A score ≤12 indicates that pain is unlikely to have a neuropathic component (< 15%), while a score of ≥19 suggests that pain is likely to have a neuropathic component (> 90%). An intermediate score (≥13, ≤18) indicates a possible neuropathic component.
Patient satisfaction | 2 and 6 weeks after surgery and 3, 6, 12, 24, 60 ,120 months after surgery
  0-10 numeric rating scale (NRS)
Post-operative nausea | first 3 days post-operative days during hospitalisation
  incidence and intensity (on a 0-10 NRS) will be evaluated. The 0-10 NRS is a valid and reliable instrument used for the self- assessment of symptoms: it consists in a single 11-point numeric scale, with 0 indicating no nausea and 10 reflecting the worst possible nausea
Post-operative opioids and analgesic drugs consumption | first 3 days post-operative days during hospitalisation
  Medication Quantification Scale (MQS) score. It is calculated for each medication by taking a consensus-based detriment weight for a given pharmacologic class and multiplying it by a score for dosage. The calculated values for each medication are then summed for a total MQS score. The score can provide a useful point measure of medication usage for any pain medication regime
Postoperative inflammatory response | preoperatively and first 3 days post-operative days during hospitalisation
  This outcome will be evaluated in terms of hematic C-Reactive Protein (CRP) and erythrocyte sedimentation rate (ESR) (the medical chart will be evaluated)
Time from surgery to first mobilization | During Hospitalization, approximately 1 days
  Time from surgery to first mobilization
Rate of frozen shoulders | 1 week post-operative during hospitalisation
  This is considered a complication occurring up to 11% and is induced by postoperative inflammatory processes that can lead to adhesive capsulitis

OTHER OUTCOMES:
Rate of serious adverse events related to steroid supplementation | 2 and 6 weeks after surgery and 3, 6, 12, 24, 60 ,120 months after surgery
  Rate of serious adverse events related to steroid supplementation
Rate of prosthetic joint infections | 2 and 6 weeks after surgery and 3, 6, 12, 24, 60 ,120 months after surgery
  Rate of prosthetic joint infections
Rate of wound infections | 2 and 6 weeks after surgery and 3, 6, 12, 24, 60 ,120 months after surgery
  Rate of wound infections
Rate of wound healing problems | 2 and 6 weeks after surgery and 3, 6, 12, 24, 60 ,120 months after surgery
  Rate of wound healing problems

CONTACTS AND LOCATIONS:
Overall Officials: Christian Candrian, Prof.Dr.med, Principal Investigator — EOC
Locations (1):
- Christian Candrian, Lugano, Switzerland

IPD SHARING:
Plan to Share IPD: No
not foreseen